CLINICAL TRIAL: NCT00406588
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study of SLV308 as Adjunct Therapy to Levodopa in Patients With Parkinson's Disease Experiencing Motor Fluctuations.
Brief Title: SLV308 for Treatment of Patients With Parkinson's Disease Experiencing Motor Fluctuations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S308.3.002; 2006-005182-20
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2008-07

CONDITIONS: Advanced Stage Parkinson's Disease
Keywords: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; pardoprunox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Levodopa (Pardoprunox)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Levodopa (Pardoprunox) — 12-42mg
  Arms: 1
Drug: Placebo Comparator — Placebo
  Arms: 2

SUMMARY:
This study is a multicenter, randomized, double blind, parallel group study of 3 months' treatment with SLV308 administered as a monotherapy in patients with advance stage PD. An open label safety extension to this study is planned as a separate protocol for patients who are willing and eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease,
* advance stage of disease,
* Modified Hoehn & Yahr stage II-IV,
* presence of a recognizable 'on' and 'off' state (motor fluctuations) and stable treatment with levodopa for at least 28 days prior to randomization

Exclusion Criteria:

* 'on-off' phenomena or 'yo-yoing' and/or an abrupt unpredictable loss of efficacy unrelated to the timing of L-DOPA administration,
* Prevalent expression of troublesome dyskinesias during 'on' time at waking hours,
* Diagnosis is unclear or a suspicion of other parkinsonian syndromes exists,
* Previous surgery for the treatment of PD

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of the maintenance period or at the early termination visit in 'off'-time as recorded in patients' home diaries. | 12 weeks

SECONDARY OUTCOMES:
Increase of 'on'-time, change from baseline in the total score of the UPDRS part 2+3, and PDQ-39 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (87):
- United States (15):
  - Site 223, Birmingham, Alabama
  - Site 220, La Jolla, California
  - Site 211, San Francisco, California
  - Site 214, Fort Lauderdale, Florida
  - Site 218, Gainsville, Florida
  - Site 213, Tampa, Florida
  - Site 219, Augusta, Georgia
  - Site 221, Chicago, Illinois
  - Site 216, Kansas City, Kansas
  - Site 224, Lexington, Kentucky
  - Site 212, East Lansing, Michigan
  - Site 217, St Louis, Missouri
  - Site 222, Durham, North Carolina
  - Site 210, Toledo, Ohio
  - Site 215, Houston, Texas
- Argentina (10):
  - Site 100, Buenos Aires
  - Site 101, Buenos Aires
  - Site 102, Buenos Aires
  - Site 103, Buenos Aires
  - Site 106, Buenos Aires
  - Site 107, Buenos Aires
  - Site 109, Buenos Aires
  - Site 105, Córdoba
  - Site 104, Mar del Plata
  - Site 108, Santa Fe
- Brazil (11):
  - Site 114, Alto da Glória
  - Site 113, Belo Horizonte
  - Site 112, Campinas
  - Site 116, Marília
  - Site 111, Porto Alegre
  - Site 118, Porto Alegre
  - Site 117, Ribeirão Preto
  - Site 119, Salvador
  - Site 110, São Paulo
  - Site 115, São Paulo
  - Site 125, São Paulo
- Bulgaria (5):
  - Site 123, Plovdiv
  - Site 120, Sofia
  - Site 121, Sofia
  - Site 122, Sofia
  - Site 124, Sofia
- Canada (10):
  - Site 136, Calgary
  - Site 137, Greenfield Park
  - Site 133, Halifax
  - Site 132, Markham
  - Site 130, Montreal
  - Site 134, Ottawa
  - Site 138, Peterborough
  - Site 135, Sainte-Anne
  - Site 139, Toronto
  - Site 131, Windsor
- Chile (4):
  - Site 140, Santiago
  - Site 141, Santiago
  - Site 143, Santiago
  - Site 142, Valdivia
- Colombia (5):
  - Site 151, Bogotá
  - Site 152, Bogotá
  - Site 153, Bogotá
  - Site 154, Bogotá
  - Site 150, Medellín
- Site 160, Riga, Latvia
- Lithuania (3):
  - Site 172, Kaunas
  - Site 170, Vilnius
  - Site 171, Vilnius
- Peru (5):
  - Site 184, Bellavista Callao
  - Site 180, Lima
  - Site 181, Lima
  - Site 182, Lima
  - Site 183, Lima
- Russia (9):
  - Site 193, Kazan'
  - Site 190, Moscow
  - Site 194, Moscow
  - Site 197, Moscow
  - Site 191, Saint Petersburg
  - Site 192, Saint Petersburg
  - Site 195, Saint Petersburg
  - Site 198, Saint Petersburg
  - Site 196, Yaroslavl
- Ukraine (9):
  - Site 204, Dnipro
  - Site 206, Kharkiv
  - Site 201, Kyiv
  - Site 202, Kyiv
  - Site 205, Lviv
  - Site 203, Poltava
  - Site 208, Simferopol
  - Site 200, Vinnitsa
  - Site 207, Zaporizhya

REFERENCES:
- [Derived] Rascol O, Bronzova J, Hauser RA, Lang AE, Sampaio C, Theeuwes A, van de Witte SV. Pardoprunox as adjunct therapy to levodopa in patients with Parkinson's disease experiencing motor fluctuations: results of a double-blind, randomized, placebo-controlled, trial. Parkinsonism Relat Disord. 2012 May;18(4):370-6. doi: 10.1016/j.parkreldis.2011.12.006. Epub 2012 Feb 7. PMID 22316635